CLINICAL TRIAL: NCT06476652
Title: Effect of Simple Simulator-based Training on Initial Performance of Novices in Ultrasound-guided Adductor Canal Block
Brief Title: Effect of Simple Simulator-based Training on Initial Performance of Novices Iultrasound-guided Adductor Canal Block
Status: Enrolling by invitation | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Teerawat Krongyut, Principal Investigator, Prince of Songkla University
Other Study IDs: REC.67-155-8-4
Record Dates: First submitted 2024-06-09; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective descriptive study is effect of simple simulator-based training on initial performance of novices in ultrasound-guided adductor canal block. The main question is Can we improve performance on simple simultor-based training ultrasound-guide adductor canal block?. We evaluate in First-year residents in Anesthesiology, Faculty of medicine, PSU.

ELIGIBILITY:
Inclusion Criteria:

* First-year anesthesiology residents in faculty of medicine, PSU

Exclusion Criteria:

* Residents with previous experience in ultrasound-guide adductor canal block

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: we choose First-year anesthesiology residents in faculty of medicine, PSU
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The efficiency of using a simple model for injecting local anesthesia through the adductor canal under ultrasound guidance assessed by Design and Validation Regional Anaesthesia Procedural skill Assessment tool | 1 year
  To study the efficiency of using a simple model for injecting local anesthesia through the adductor canal under ultrasound by 1st year anesthesia residentassessed by Design and Validation Regional Anaesthesia Procedural skill Assessment tool

SECONDARY OUTCOMES:
satisfaction and confidence in teaching assessed by pre- and post-test, satisfaction questions | 1 year
  To study satisfaction and confidence in teaching by using a simple simulator for injecting regional anesthesia through the adductor canal under ultrasound guidance by anesthesiology resident with no prior experience assessed by pre- and post-test, satisfaction question

CONTACTS AND LOCATIONS:
Overall Officials: Teerawat Krongyut, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand